CLINICAL TRIAL: NCT01343524
Title: Changes in Lung Function Based on Differences in Spirometry Equipment Used in Children With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Ran Anbar, Professor, State University of New York - Upstate Medical University
Other Study IDs: 5891
Record Dates: First submitted 2011-02-14; First posted 2011-04-28 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; spirometry; PFT's; pulmonary function test
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- all subjects: all subjects who are enrolled in an industry-sponsored study that utilizes a sponsor-supplied spirometer.

SUMMARY:
The investigators' Upstate Cystic fibrosis (CF) Care Center is very active in research. For example, in 2009, 68 of our 135 pediatric patients have been participating in 16 clinical trials. Sponsors often provide their study sites with spirometers to use for PFTs. These machines are meant to provide uniform PFTs results for studies, which include measurement of FEV1 values. In 2009, among the 52 patients at our Center who are 6-12 years old, 20 (38%) have been in studies with sponsor-provided spirometers. Among the 32 patients ages 13-17 years, 13 (40%) have been in studies with sponsor-provided spirometers. Anecdotally, the investigators have noted that FEV1 results obtained during clinical trials for our patients appear to be lower than those of our patients' usual values, especially with younger children. The investigators hypothesize that the apparent difference in PFT results might be related to the different incentives (if any) provided by study PFT equipment. Further, if this difference exists, the investigators believe that this may account for the apparent average decline in the lung function results of our patients over the recent years, given the large proportion of our patients who participate in clinical trials. Finally, the investigators hypothesize that younger children may be more affected by the difference in incentives than older ones.

The purpose of this study is to collect an additional set of Pulmonary Function Tests (PFTs) using our regular clinic equipment, on all study subjects following their study PFTs if these are done with sponsor-provided equipment. The investigators will compare the results from both types of machines and report regarding differences identified.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is an autosomal recessive genetic disease, characterized by pulmonary and sinus disease, gastrointestinal and reproductive tract dysfunction. CF patients suffer from chronic repeated cycles of pulmonary bacterial infection, pulmonary exacerbations and chronic lung function decline, which often lead to premature death. Although improved treatment of lung disease has increased survival, the median predicted age for survival is only 37.2 years in the United States (US) (CFF Annual Data Report, 2008) and patients continue to have significant morbidity, including hospitalizations (Ramsey, 1996).

Pulmonary Function Tests (PFTs) are used to measure and track lung health of patients with CF. Performing a PFT takes practice and requires patients to perform certain breathing maneuvers consistently. Infants and young children cannot be tested using spirometers. The investigators start PFT training with our patients after they reach 4 years of age. It may take several months to a few years for useful, consistent and interpretable PFTs to be obtained. According to standards developed by the American Thoracic Society, children must be able to breathe in very deeply, exhale fast and hard, and continue exhaling for several seconds. Children also must perform these maneuvers in a repeatable manner. (Ferris, 1978 ). Recent software programs have been developed to encourage and assist children in completing the breathing maneuvers. Videogame-like graphics respond to children's efforts. Children can often choose which "game" to play, such as, "Blow out the candles."

PFT results have taken on greater importance as new therapies are tested and evaluated. One component of the PFT is the FEV1 value (the amount of air exhaled in one second). Physicians, families and patients keep track of the FEV1 values and decreases are investigated carefully and addressed with treatment modification, if necessary. Many industry-sponsored and CF Foundation-sponsored protocols use FEV1 values in their exclusion and inclusion criteria for studies involving patients with CF. FEV1 is used to judge the efficacy of most investigational treatments. (In many studies, change in FEV1 is the only primary endpoint measured.)

Almost all of our patients with CF participate in the national CF Foundation (CFF)-sponsored CF Registry. Detailed clinical information is collected through the Registry and published each year in the CFF Annual Data Report and online, from which some of the information is accessible to the public. The Data Report is meant to be one way to compare outcomes at different CF Centers. Also, it is used locally to identify areas that need further improvement. In the recently published 2008 Data Report, the average FEV1 values for patients at our Center ages 6-12 years had decreased significantly from last year. This continues a trend the investigators have seen over the past 5 years, despite no apparent change in the treatment protocols at our Center. Nationally, FEV1 values for patients in this age range have stayed the same. This apparent local decrease was quite troubling to our Center staff and became a recent focus of our Quality Improvement efforts.

Our Upstate CF Care Center is very active in research. For example, in 2009, 68 of our 135 pediatric patients have been participating in 16 clinical trials. Sponsors often provide their study sites with spirometers to use for PFTs. These machines are meant to provide uniform PFTs results for studies, which include measurement of FEV1 values. In 2009, among the 52 patients at our Center who are 6-12 years old, 20 (38%) have been in studies with sponsor-provided spirometers. Among the 32 patients ages 13-17 years, 13 (40%) have been in studies with sponsor-provided spirometers. Anecdotally, the investigators have noted that FEV1 results obtained during clinical trials for our patients appear to be lower than those of our patients' usual values, especially with younger children. The investigators hypothesize that the apparent difference in PFT results might be related to the different incentives (if any) provided by study PFT equipment. Further, if this difference exists, the investigators believe that this may account for the apparent average decline in the lung function results of our patients over the recent years, given the large proportion of our patients who participate in clinical trials. Finally, the investigators hypothesize that younger children may be more affected by the difference in incentives than older ones.

The purpose of this study is to collect an additional set of PFTs using our regular clinic equipment, on all study subjects following their study PFTs if these are done with sponsor-provided equipment. The investigators will compare the results from both types of machines and report regarding differences identified.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cystic fibrosis (CF)
* Enrolled in an industry-sponsored CF study that requires use of a sponsor-supplied spirometer
* Capable of performing Pulmonary Function Test (PFT)
* Less than 22 years old

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will include CF patients enrolled in studies that require PFTs using study-provided spirometers. Any patient less than 22 years old, capable of performing PFTs for research studies, will be offered this study as well.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Comparison of Pulmonary Function (FVC, FEV1) on 2 different spirometers | 1/1/2009-12/31/2010
  We plan to compare a subject's FVC and FEV1 values obtained on the same day, within 15 minutes of each other, done on our familiar clinic spirometer and on the less familiar study spirometer. ASSESSMENT OF EFFICACY
  Primary Efficacy Parameters
  • FEV1 (L)
  Statistics
  We will compare the average FEV1 for study and non-study PFTs by using a Student's t-test. Additionally, we will compare the difference in PFT's among children in the 6-12 year old age groups, with those in the 13-17 year old age group (which is the same age breakdown that is reported in the CF Foundation Data Report.)

CONTACTS AND LOCATIONS:
Overall Officials: Ran D Anbar, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

REFERENCES:
- [Background] Cystic Fibrosis Foundation 2008 Annual Data Report; http://www.cff.org/UploadedFiles/aboutCFFoundation/Publications/AnnualReport/Final%202 006%20Annual%20Report.pdf.
- [Background] Ferris BG. Epidemiology Standardization Project (American Thoracic Society). Am Rev Respir Dis. 1978 Dec;118(6 Pt 2):1-120. No abstract available. PMID 742764
- [Background] Ramsey BW. Management of pulmonary disease in patients with cystic fibrosis. N Engl J Med. 1996 Jul 18;335(3):179-88. doi: 10.1056/NEJM199607183350307. No abstract available. PMID 8657217